CLINICAL TRIAL: NCT00865228
Title: A Double-blind, Randomized Study to Evaluate the Efficacy and Safety of Lapaquistat Acetate 100 mg in the Morning vs Lapaquistat Acetate 100 mg in the Evening vs Lapaquistat Acetate 50 mg Twice Daily vs Placebo in Subjects With Hypercholesterolemia
Brief Title: Efficacy of Lapaquistat Acetate in Subjects With Hypercholesterolemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Overall profile of the compound does not offer significant clinical advantage to patients over currently available lipid lowering agents
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-475_201; U1111-1122-8404 (Registry Identifier: WHO)
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Dyslipidemia; High Cholesterol; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lapaquistat Acetate 100 mg QD (morning) (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Lapaquistat Acetate 100 mg QD (evening) (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Lapaquistat Acetate 50 mg BID (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lapaquistat acetate — Lapaquistat acetate 100 mg, tablets, orally, once daily in the morning and Lapaquistat acetate placebo-matching tablets, orally, once daily in the evening for up to six weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD (morning)
Drug: Lapaquistat acetate — Lapaquistat acetate placebo-matching tablets, orally, once daily in the morning and Lapaquistat acetate 100 mg, tablets, orally, once daily in the evening for up to six weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD (evening)
Drug: Lapaquistat acetate — Lapaquistat acetate 50 mg, tablets, orally, once daily in the morning and Lapaquistat acetate 50 mg, tablets, orally, once daily in the evening for up to six weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 50 mg BID
Drug: Placebo — Lapaquistat acetate placebo-matching tablets, orally, once daily in the morning and Lapaquistat acetate placebo-matching tablets, orally, once daily in the evening for up to six weeks.
  Arms: Placebo BID

SUMMARY:
The purpose of this study is to determine the role of time of dosing on the lipid-lowering effects of lapaquistat acetate, once daily (QD) or twice daily (BID), in subjects with hypercholesterolemia.

DETAILED DESCRIPTION:
Dyslipidemias are a group of metabolic disorders produced by raised concentrations of lipoproteins, especially low-density lipoprotein cholesterol the lipoprotein that transports endogenous cholesterol from the liver to the peripheral tissues. Increased cholesterol and triglyceride levels lead to an increased risk of arteriosclerosis, the underlying cause of heart attack, strokes and peripheral vascular disease. Despite changes in lifestyle and the availability of potent lipid-lowering agents, cardiovascular disease continues to be the major cause of death in Western Europe and North America.

Lapaquistat acetate is being developed by Takeda for the treatment of hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use a medically accepted means of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Has prior to Randomization a mean low-density lipoprotein cholesterol greater than or equal to 130 mg/dL and less than or equal to 220 mg/dL for 2 consecutive samples.
* Has prior to Randomization mean triglycerides less than 400 mg/dL for 2 consecutive samples.
* Is willing and able to comply with a standardized, therapeutic lifestyle change diet or equivalent.

Exclusion Criteria:

* Has an alanine aminotransferase or aspartate aminotransferase level greater than 2 times the upper limit of normal during the screening period.
* Has a serum creatinine greater than133 mmol/L during the screening period.
* Has a creatine phosphokinase greater than 3 times the upper limit of normal, identified during the screening period.
* Has active liver disease or jaundice.
* Has a history of cancer that has been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, unstable angina, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdomin al aorticaneurysm, coronary angioplasty, coronary or peripheral arterial surgery or multiple risk factors that confer a 10-year risk for cardiovascular disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen, or antibody to hepatitis C virus, as determined by medical history and/or subject's verbal report.
* Has a positive human immunodeficiency virus status or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Has received any investigational compound within 30 days prior to screening Visit 1, or is currently participating in another investigational study.
* Has received lapaquistat acetate in a previous clinical study or as a therapeutic agent.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the specialized diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia.
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension despite treatment at Screening Visit 1.
* Has had inflammatory bowel or any other malabsorption syndrome or has had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or alcohol abuse within the past 2 years.
* Has stage I squamous cell carcinoma of the skin.
* Has type 1 or type 2 diabetes mellitus.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Fluvastatin
  * Lovastatin
  * bile acid sequestrants (eg, cholestyramine)
  * intestinal cholesterol uptake inhibitors (eg, ezetimibe)
  * Fibrates (eg, fenofibrate, gemfibrozil)
  * Niacin
  * Cholestin
  * red yeast rice
  * fish oils
  * plant sterols and stanols
  * orlistat
  * sibutramine
  * isotretinoin
  * tacrolimus
  * Probucol
  * Systemic corticosteroids and androgens
  * Potent CYP3A4 inhibitors
  * Cyclosporine
  * Erythromycin
  * Clarithromycin
  * Telithromycin
  * human immunodeficiency virus protease inhibitors
  * amiodarone
  * diltiazem
  * verapamil
  * nefazodone
  * grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in the Fasting Plasma Low-Density Lipoprotein Cholesterol concentration | Week 6

SECONDARY OUTCOMES:
Change from Baseline in Total Cholesterol | Week 6
Percent change from Baseline in apolipoprotein B | Week 6
Percent change from Baseline in apolipoprotein A1 | Week 6
Change from Baseline in Triglycerides | Week 6
Percent change from Baseline in High-Density Lipoprotein Cholesterol | Week 6
Percent change from Baseline in Very Low-Density Lipoprotein Cholesterol | Week 6
Percent change from Baseline in non- High-Density Lipoprotein Cholesterol | Week 6
Percent change from Baseline in derived ratio of Low-Density Lipoprotein Cholesterol / High-Density Lipoprotein Cholesterol | Week 6
Percent change from Baseline in derived ratio of Total Cholesterol / High-Density Lipoprotein Cholesterol | Week 6
Percent change from Baseline in derived ratio of apolipoprotein B / apolipoprotein A1 | Week 6
Change from Baseline in high sensitivity C-Reactive Protein. | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Science, Study Director — Takeda
Locations (22):
- United States (22):
  - Long Beach, California
  - Sacramento, California
  - San Diego, California
  - Hollywood, Florida
  - Jacksonville, Florida
  - New Port Richey, Florida
  - Chicago, Illinois
  - Wichita, Kansas
  - Louisville, Kentucky
  - Margate City, New Jersey
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Medford, Oregon
  - Perkasie, Pennsylvania
  - Sellerville, Pennsylvania
  - Bristol, Tennessee
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin